CLINICAL TRIAL: NCT04556396
Title: Intraoperative Cone-beam CT for Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Kristin Baldea, MD, Assistant Professor Of Urology, Loyola University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212740
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Nephrolithiasis
Keywords: percutaneous nephrolithotomy; cone beam CT
MeSH Terms: conditions — Nephrolithiasis | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Intervention Model Description: Patients are assigned to receive intraoperative cone beam CT if enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention arm (Experimental): This arm will receive cone beam CT to perform an abdomen-pelvis CT scan immediately following initial percutaneous nephrolithotomy, before the patient emerges from general anesthesia, to allow the surgeon to determine whether additional work is needed or whether the procedure can be concluded without requiring further imaging or future interventions.
  Interventions: Diagnostic Test: Cone beam CT
- Retrospective arm (No Intervention): This arm will contain a retrospective cohort of patients who underwent surgery prior to the enrollment of the intervention arm. These patients received the standard of care, namely helical CT postoperative day one.

INTERVENTIONS:
Diagnostic Test: Cone beam CT — On-table CT scan in the operating room to determine residual kidney stone burden at end of procedure
  Other Names: O-arm; Intraoperative CT
  Arms: Intervention arm

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is a first-line treatment for kidney stones >2cm. Frequently, patients require multiple procedures to address their stone burden. The decision to proceed with a second-look procedure is based on follow-up CT imaging, which is obtained postoperatively. In this study, we propose the use of a portable CT scan technology to obtain follow-up imaging while the patient is still under anesthesia for the initial procedure. The goal of this study is to determine whether this allows the surgeon to identify residual fragments and render the patient stone-free within a single anesthetic event.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is considered a first-line management option for kidney stones larger than two centimeters. Unfortunately, because of the large stone burden, up to 70% of these patients are left with residual stone fragments after their initial PCNL. Additionally, an estimated 20% to 60% of such patients ultimately require further interventions due to residual stone fragments. The need for a subsequent procedure is determined by postoperative abdominal computed tomography (CT) imaging, which is routinely performed on the first postoperative day at this institution. The decision to proceed with a second procedure is based on findings from this postoperative CT scan.

Cone-beam CT (CBCT) is a novel portable imaging technique that can allow cross-sectional imaging to be obtained intraoperatively, rather than post-operatively. Incorporating this modality would allow the surgeon to determine whether the procedure should be continued, in the event of residual fragments, or if it can be safely concluded. This would obviate the need for dedicated postoperative CT scans and, more importantly, reduce the need for subsequent procedures and consequently decrease the patient's length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years old
2. Scheduled for percutaneous nephrolithotomy with stone fragmentation (laser/ultrasonic/mechanical)
3. For the prospective intervention arm, willingness to consent to participate in the study

Exclusion Criteria:

1. Patients whose habitus does not allow for the use of the cone beam CT machine
2. Patients whose stones only reside within the mid or distal ureter(s) and thus would not be easily imaged with cone beam CT
3. Patients who have had lithotripsy on their renal unit within the prior 90 days
4. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin G Baldea, MD, Principal Investigator — Attending Physician
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearle MS, Watamull LM, Mullican MA. Sensitivity of noncontrast helical computerized tomography and plain film radiography compared to flexible nephroscopy for detecting residual fragments after percutaneous nephrostolithotomy. J Urol. 1999 Jul;162(1):23-6. doi: 10.1097/00005392-199907000-00006. PMID 10379731
- [Background] Nevo A, Holland R, Schreter E, Gilad R, Baniel J, Cohen A, Lifshitz DA. How Reliable Is the Intraoperative Assessment of Residual Fragments During Percutaneous Nephrolithotomy? A Prospective Study. J Endourol. 2018 Jun;32(6):471-475. doi: 10.1089/end.2018.0005. Epub 2018 Mar 23. PMID 29466870
- [Background] Roy OP, Angle JF, Jenkins AD, Schenkman NS. Cone beam computed tomography for percutaneous nephrolithotomy: initial evaluation of a new technology. J Endourol. 2012 Jul;26(7):814-8. doi: 10.1089/end.2011.0478. Epub 2012 Mar 26. PMID 22296493
- [Background] Pitteloud N, Gamulin A, Barea C, Damet J, Racloz G, Sans-Merce M. Radiation exposure using the O-arm(R) surgical imaging system. Eur Spine J. 2017 Mar;26(3):651-657. doi: 10.1007/s00586-016-4773-0. Epub 2016 Sep 21. PMID 27652675
- [Derived] Patel PM, Kandabarow AM, Chuang E, McKenzie K, Druck A, Seffren C, Blanco-Martinez E, Capoccia E, Farooq AV, Branch J, Turk TMT, Baldea KG. Using Intraoperative Portable CT Scan to Minimize Reintervention Rates in Percutaneous Nephrolithotomy: A Prospective Trial. J Endourol. 2022 Oct;36(10):1382-1387. doi: 10.1089/end.2022.0049. Epub 2022 Sep 13. PMID 35620899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Retrospective Arm
Started | 60 | 174
Completed | 60 | 174
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Retrospective Arm | Total
Number analyzed (Participants) | 60 | 174 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15) | 57 (15) | 57.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 88 | 125
  Male | 23 | 86 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 145 | 191
  Black | 5 | 12 | 17
  Other | 3 | 11 | 14
  Unknown | 2 | 1 | 3
  Asian | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 6 | 21 | 27
  Ethnicity: Non-Hispanic | 54 | 151 | 205
  Ethnicity: Unknown | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 60 | 174 | 234

OUTCOME MEASURES:

1. Primary Outcome: "Second Look" Rate
Description: The percentage of patients requiring subsequent surgical intervention to remove residual stones
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Retrospective Arm
Number analyzed (Participants) | 60 | 174
Participants
  Reintervention | 4 | 56
  No Reintervention | 56 | 118
Statistical Analysis 1: Comparison: Intervention Arm vs Retrospective Arm; Test type: Superiority; p < 0.01, Chi-squared; Odds Ratio (OR) = 0.2, 95% CI 2-sided [0.1 to 0.4]

2. Secondary Outcome: Hospital Length of Stay
Description: The average length of inpatient hospital stay in days
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Arm | Retrospective Arm
Number analyzed (Participants) | 60 | 174
Days | 2.3 (1.5) | 3.5 (2.5)

3. Secondary Outcome: Surgical Complication Rate
Description: The percentage of patients experiencing Clavien-Dindo Grade III-V complications (major) related to the patients' surgery.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Retrospective Arm
Number analyzed (Participants) | 60 | 174
Participants | 2 | 17

4. Secondary Outcome: "Stone Free" Rate
Description: The percentage of patients who are rendered without residual kidney stone burden after their surgery based on CT scan
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Retrospective Arm
Number analyzed (Participants) | 60 | 174
Participants | 49 | 63

5. Secondary Outcome: Reobstruction Rate
Description: The percentage of patients who presented with symptoms of renal obstruction following their surgery
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Retrospective Arm
Number analyzed (Participants) | 60 | 174
Participants | 11 | 26

ADVERSE EVENTS:
Time Frame: Time frame used to assess outcomes and adverse events was 90 days post index procedure
Arm/Group | Intervention Arm | Retrospective Arm
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/174
Other Adverse Events (participants affected / at risk) | 0/60 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04556396/Prot_SAP_000.pdf